CLINICAL TRIAL: NCT04742829
Title: Evaluation of the Effect of a Therapy With INTRAVIT® Tablets on Retinal Edema, Retinal Sensitivity and Visual Acuity in the Course of Diabetic Retinopathy
Brief Title: Effects of a Therapy With INTRAVIT® Tablets in Patients With Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09/2020
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; macula edema; microperimetry; curcumin; artemisin; piperine; bromelain
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Observational study, open, controlled between homogeneous groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP 1 (Experimental): Patients treated with INTRAVIT® tablets
  Interventions: Dietary Supplement: INTRAVIT ®
- GROUP 2 (No Intervention): patients who will not take any medical therapy to overlap with the activity described for INTRAVIT® tablets.

INTERVENTIONS:
Dietary Supplement: INTRAVIT ® — 2 tablets per day morning and evening before meals
  Arms: GROUP 1

SUMMARY:
Evaluation of the effect of a therapy with INTRAVIT® tablets, on retinal edema considering also the central retinal sensitivity (Microperimetry) and the visual acuity in course of diabetic retinopathy.

DETAILED DESCRIPTION:
Retinal edema is an abnormal accumulation of fluids in the retina, is a complication of certain eye diseases such as diabetic retinopathy, exudative macular degeneration, surgical or para - surgical practices and trauma. The main factors involved in the formation of retinal edema are due to structural alterations of blood vessels, formation of neovessels and phlogistic phenomena. INTRAVIT® is a product based on extracts of Artemisia, Turmeric, Pineapple and Black Pepper, formulated in a targeted way to support the treatment of retinal edema and treatments with intravitreal injections. Artemisia (artemisinin and its derivatives) has proven to be able to counteract the activity of VEGF, VEGFR, metal protein (MM2 and MMP9) and integrins αvβ3, all factors involved in the angiogenetic process. Turmeric (curcumin) has been shown to be able to counteract the phlogistic processes in various districts in addition to acting on the reduction of angiogenesis. The Pineapple (Bromelain) for its proteolytic activity has been able to favor the resorption of the edema and the reduction of the phlogistic phenomena. Black pepper (piperine) has proven to be able to counteract the phlogistic processes and encourage the bioavailability of some natural extracts such as curcumin.

The purpose of the study is to evaluate the effect of a therapy with INTRAVIT® tablets, on retinal edema considering also the central retinal sensitivity (Microperimetry) and visual acuity in the course of diabetic retinopathy. Diabetic patients with mild non-proliferant diabetic retinopathy (at an early stage) with macular edema will be enlisted. 40 patients, of which 20 will be treated with INTRAVIT® tablets (2 tablets per day morning and evening before meals), and 20 who will not take any medical therapy to overlap with the activity described for INTRAVIT® (control group). Patients covered by the inclusion criteria will undergo, before the start of treatment, a full eye examination and OCT (optical coherence tomography) for the measurement of foveal thickness. Based on the preordered randomization scheme they will be assigned to Group 1 or Group 2 (control group). Patients will undergo a first examination at the time of recruitment (T0), and subsequent visits (T1-T2) will fall to 3 and 6 months.The data collection sheet will report all adverse effects potentially attributable to the administration of the food supplement INTRAVIT® tablets.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type I and type II patients;
* Between 20 and 70 years of age;
* Age of diabetes not less than 5 years and not more than 15;
* Mild non-proliferating diabetic retinopathy, limited to the presence of some microaneurysms;
* Patients in diabetic compensation;
* Visual acuity 5/10 natural or correct;
* Patients even if hypertensive, with or without anti-hypertensive therapy in place, provided they are compensated;
* Patients with good visualization of the ocular fundus.

Exclusion Criteria:

* Patients with concurrent eye diseases outside diabetic retinopathy;
* Patients with less than natural or correct 5/10 visual acuity;
* Patients treated with other vasoprotective and antioxidant preparations or having taken them in the last month;
* Patients with significant systemic or metabolic diseases, except diabetes;
* Patients with unbalanced Diabetes disorder;
* Patients undergoing laser treatment or eye surgery (e.g. cataract);
* Patients who take or should take, during the observation period, preparations for direct or indirect activity on the retina of the type that can be superimposed on INTRAVIT ®.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-08 (Estimated); Study Completion 2021-03-08 (Estimated)

PRIMARY OUTCOMES:
number of participants with signs of improvement/worsening of diabetic retinopathy | 6 months
  report presence/absence of signs with Yes/NO relative to: microaneurysms, haemorrhages, soft exudates, hard exudates, venous beading, IRMA, new vessels on optical discs, new vessels outside the optical discs, cystoid edema, capillary occlusions, degenerative alterations and vein size.
number of participants in a certain stage of diabetic retinopathy according to the ETDRS modified AAO 2003 | 6 months
  careful evaluation of funduscopic signs (e.g exudates, neovases, micronaneurysms) to be able to stadiate patients
number of patients with improved/worsened visual acuity | 6 months
  visual acuity measurement with ETDRS boards. The number of letters seen by the patient at each check-up visit will be noted.
number of patients with improved/worsened macular edema | 6 months
  Foveal thickness (measured with Optical Coherence Tomography) at each check-up visit will be noted.

SECONDARY OUTCOMES:
number of patients with improved/worsened blood parameters related to diabetes | 6 months
  blood sugar (mg/dl) using a rapid glucose test at each check-up visit will be noted and glycated hemoglobin (%) will be assesed with venous blood sampling at the beginning of the study and at 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Molise, Campobasso, Italy

REFERENCES:
- [Result] Wang W, Lo ACY. Diabetic Retinopathy: Pathophysiology and Treatments. Int J Mol Sci. 2018 Jun 20;19(6):1816. doi: 10.3390/ijms19061816. PMID 29925789
- [Result] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Result] Yang F, Yu J, Ke F, Lan M, Li D, Tan K, Ling J, Wang Y, Wu K, Li D. Curcumin Alleviates Diabetic Retinopathy in Experimental Diabetic Rats. Ophthalmic Res. 2018;60(1):43-54. doi: 10.1159/000486574. Epub 2018 Mar 29. PMID 29597206
- [Result] Radomska-Lesniewska DM, Osiecka-Iwan A, Hyc A, Gozdz A, Dabrowska AM, Skopinski P. Therapeutic potential of curcumin in eye diseases. Cent Eur J Immunol. 2019;44(2):181-189. doi: 10.5114/ceji.2019.87070. Epub 2019 Jul 30. PMID 31530988
- [Result] Mohr T, Desser L. Plant proteolytic enzyme papain abrogates angiogenic activation of human umbilical vein endothelial cells (HUVEC) in vitro. BMC Complement Altern Med. 2013 Sep 21;13:231. doi: 10.1186/1472-6882-13-231. PMID 24053149
- [Result] Al-Malki AL. Shikimic acid from Artemisia absinthium inhibits protein glycation in diabetic rats. Int J Biol Macromol. 2019 Feb 1;122:1212-1216. doi: 10.1016/j.ijbiomac.2018.09.072. Epub 2018 Sep 15. PMID 30227208
- [Result] Kumar S, Sharma S, Vasudeva N. Screening of antidiabetic and antihyperlipidemic potential of oil from Piper longum and piperine with their possible mechanism. Expert Opin Pharmacother. 2013 Sep;14(13):1723-36. doi: 10.1517/14656566.2013.815725. Epub 2013 Jul 23. PMID 23875561
- [Result] Pescosolido N, Giannotti R, Plateroti AM, Pascarella A, Nebbioso M. Curcumin: therapeutical potential in ophthalmology. Planta Med. 2014 Mar;80(4):249-54. doi: 10.1055/s-0033-1351074. Epub 2013 Dec 9. PMID 24323538
- [Result] Maugeri A, Mazzone MG, Giuliano F, Vinciguerra M, Basile G, Barchitta M, Agodi A. Curcumin Modulates DNA Methyltransferase Functions in a Cellular Model of Diabetic Retinopathy. Oxid Med Cell Longev. 2018 Jul 2;2018:5407482. doi: 10.1155/2018/5407482. eCollection 2018. PMID 30057682
- [Result] Wilkinson CP, Ferris FL 3rd, Klein RE, Lee PP, Agardh CD, Davis M, Dills D, Kampik A, Pararajasegaram R, Verdaguer JT; Global Diabetic Retinopathy Project Group. Proposed international clinical diabetic retinopathy and diabetic macular edema disease severity scales. Ophthalmology. 2003 Sep;110(9):1677-82. doi: 10.1016/S0161-6420(03)00475-5. PMID 13129861